CLINICAL TRIAL: NCT00788021
Title: Characterization of the Impact of Chronic Immunosuppressive Regimens on Protective Immunity Over Time in Renal Transplant Recipients
Brief Title: Protective Immunity Project 01
Acronym: PIP-01
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Christian P Larsen, MD, PhD, Chairman, Dept of Surgery, Emory University
Other Study IDs: IRB00000709; PIP-01 (Other: Other)
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Kidney Transplantation; Immunity; Immunosuppression
Keywords: Transplant; Immunity; Immunosuppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, PBMCs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Tacrolimus: Recipients of deceased or living donor renal transplant maintained on immunosuppressive regimen utilizing tacrolimus
- Sirolimus: Recipients of deceased or living donor renal transplants maintained on immunosuppressive regimen using sirolimus
- Healthy controls: Age, race and gender-matched individuals not on immunosuppressive regimens. Whenever possible an transplant recipient's donor may be recruited to serve as healthy control

SUMMARY:
Patients who undergo kidney transplant must take medications to prevent organ rejection. There are standard immunosuppressant medications such as prednisone, tacrolimus (Prograf), mycophenolate mofetil(Cellcept) or sirolimus (Rapamune) that are given to patients to prevent rejection. It is well known that patients on immunosuppressant medications are at increased risk from viral infections, such as influenza. However, it is not well understood how immunosuppressive medications may uniquely affect the immune response to infection. This study will determine whether there are unique differences in the effects on the immune system by these different immunosuppressive medications, particularly differences between tacrolimus and sirolimus.

DETAILED DESCRIPTION:
While the benefits of transplantation to society are substantial, the ever-growing population of immunosuppressed recipients poses a unique challenge in development of immunization and containment strategies to protect the population from communicable pathogens and weaponized infectious agents. The immunosuppressive regimens that have allowed the emergence of successful transplant therapy not only inhibit T cell-dependent rejection but also cause systemic immunosuppression, which attenuates the response to vaccines in general and precludes the use of live attenuated vaccines. To date, there has been relatively little detailed systematic study of the immune alterations that accompany either the short- or long-term immunosuppressive regimens used in clinical organ transplantation. Despite the recent development of increasingly effective, but also increasingly complex, regimens using drugs with very distinct molecular targets, current policies on vaccination of transplant recipients are generic and remain based on old concepts rather than on any new understanding of the cellular and molecular effects of these therapies on the human immune system. This proposal seeks to improve our understanding of the biological mechanisms that underlie the distinct immunosuppressive regimens in practice today (calcineurin-inhibitor, or CNI, and sirolimus-based regimens) and in emerging regimens that employ agents with novel mechanisms of action, such as the CD28 costimulation blockers, and/or JAK3 kinase inhibitors. Such knowledge will be critical to strategies for enhancing desirable immune responses while not precipitating rejection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 and 59 years of age
2. Patients capable of understanding the purposes and risks of the study, who can give written informed consent and who are willing to participate in and comply with the study.
3. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment and must not be breast-feeding.

Exclusion Criteria:

1. Patients with any prior organ transplant or multi-organ transplant recipients
2. Patients that require induction immunosuppression beyond the immunosuppressive regimen proposed in this study. For example, patients that receive anti-lymphocyte antibody therapy or plasmapheresis as a result of pre-formed immunologic reactivity to the transplanted organ.
3. Patients with evidence of an active systemic infection requiring the continued use of antibiotics, evidence of an HIV infection, or the presence of a chronic active hepatitis B or C.
4. Patients with history of malignancy in the last 5 years (except successfully treated localized non-melanotic skin cancer)
5. Patients with severe anemia (hemoglobin < 8 g/dL), leukopenia (WBC < 3000/mm3). -

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing deceased or living donor renal transplant
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2006-09; Primary Completion 2011-01 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To determine the effects of chronic immunosuppressive therapies on adaptive immunity | 2 years
To determine the effects of chronic immunosuppressive therapies on innate immunity, dendritic cell phenotype and function and TLR signaling | 2 years
To define the transcriptional signatures associated with specific immunosuppressive regimens | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian P. Larsen, MD, DPhil, Principal Investigator — Emory University; Kenneth E. Kokko, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States